CLINICAL TRIAL: NCT04793100
Title: Spontaneous Retinal Artery Pulses (SPARs) as a Prognostic Determinant of Central Retinal Vein Occlusions (CRVO) in Patients With or Without Intravitreal Aflibercept Injections
Acronym: PULSOV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MMT_2020_33
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Central Retinal Vein Occlusion
Keywords: Central Retinal Vein Occlusion; Spontaneous retinal artery pulsation
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Follow-up for 1 year (Experimental)
  Interventions: Other: Ophthalmologic exam at inclusion and 12 months after CRVO; Drug: Treatment standardization with aflibercept

INTERVENTIONS:
Other: Ophthalmologic exam at inclusion and 12 months after CRVO — As part of routine care : OCT-B (Optical coherence tomography-B), OCT-angiography (Optical coherence tomography and fluorescein angiography after pupillary dilatation (at inclusion only)
  Added by the study :
  * Assessment of best corrected visual acuity in letters read and validated using the ETDRS scale ;
  * The shooting of a 10 second infrared movie by the Heidelberg Spectralis device centered on the head of the optic nerve (at inclusion only)
  * A measurement of the eye tension with an air tonometer (at inclusion only)
  * A blood pressure measurement (diastolic and systolic) and pulse measurement (at inclusion only)
  * A color retinophotography (Optos) with autofluorescence images
  * A color Doppler ultrasound of the optic nerve of both eyes will be performed, for patients treated at the Foundation A de Rothschild Hospital only.
Drug: Treatment standardization with aflibercept — For patients requiring intravitreal injection

SUMMARY:
Central retinal vein occlusion (CRVO) is the second most common retinal vascular disease after diabetic retinopathy. It induces circulatory slowdown and blood stasis, which can appear as retinal hemorrhages. CRVO has been classically separated into two clinical forms: ischemic CVRO (possibly associated with cotton wool spots) and non-ischemic CRVO, the former being considered the most serious due to neovascular complications. More recently, a new classification has been suggested by Pierru et al. distinguishing two types of CRVO: type A characterized by low acute blood flow and type B with a slower onset. Type A is particularly associated with younger age, the presence of acute paracentral middle maculopathy, concomitant cilioretinal artery occlusion, and/or pulsatile arterial filling. Type B is more likely to occur in elderly patients, usually with high blood pressure, and multiple hemorrhages are frequently found on fundus examination.

A retrospective study had shown a slight difference in favor of pulsatile CRVO in terms of the number of intravitreal anti-angiogenic injections required to treat macular edema and visual acuity changes. However, no statistically significant difference was observed.

The objective of this study is to prospectively investigate whether spontaneous retinal artery pulses (SPARs) in patients with type A or B CRVO can be considered as a prognostic factor for the evolution of CRVO.

DETAILED DESCRIPTION:
In order to be able to interpret the results on a homogeneous population, given that several molecules have marketing authorization for the management of macular edema following a CRVO, the therapeutic management will be standardized by the use of aflibercept for patients requiring intravitreal injection, aflibercept being the most widely referenced treatment currently used in the participating centers.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CRVO, with or without macular edema.
* Onset of symptoms in the previous month (maximum 30 days prior to inclusion)
* Naive of intravitreal injection and intravitreal corticosteroid implant
* If woman of childbearing age: commitment to effective contraception during treatment with aflibercept and for at least 3 months after the last intravitreal injection of aflibercept

Exclusion Criteria:

* Pregnant or breastfeeding woman
* History of stroke or myocardial infarction in the last 3 months
* Retinal detachment or untreated retinal dehiscence
* Opacity of ocular media
* Amblyopia
* Diabetic retinopathy
* Macular edema of a different etiology than CRVO
* Active or suspected ocular or periocular infection
* Severe intraocular inflammation
* Hypersensitivity to EYLEA® : to the active substance (aflibercept) or to one of the excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-03-17 (Actual)

PRIMARY OUTCOMES:
Change in visual acuity between inclusion and visit at one year compared between patients with SPARs versus without SPARs | At inclusion and 12 months after CRVO
  Evolution of best corrected visual acuity on ETDRS scale (Early treatment diabetic retinopathy study scale) in letters read and validated Infrared movies will be made at inclusion from the Heidelberg Spectralis device. Two ophthalmologists blinded to each other will view the films. The arterial pulses are visualized at the optic disc site in the form of pulse-dependent beats of the arterial walls. For each movie each ophthalmologist will give his assessment: SPARs+ or SPARs-. In case of discrepancy, a third ophthalmological opinion will be requested.

CONTACTS AND LOCATIONS:
Overall Officials: Martine MAUGET FAYSSE, MD, Principal Investigator — Hôpital Fondation A. de Rothschild
Locations (3):
- France (3):
  - Centre Pôle Vision du Val d'ouest, Lyon, Écully
  - Hôpital Fondation A. de Rothschuld, Paris
  - Centre médical et chirurgical de la rétine Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No